CLINICAL TRIAL: NCT07287371
Title: Randomized Trial of Sucrosomial Iron Vs Intravenous Iron for Preoperative Anemia (RSIVI)
Brief Title: Sucrosomial Vs Intravenous Iron for Preoperative Anemia
Acronym: RSIVI
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Pharmanutra S.p.a. (Industry)
Responsible Party: Principal Investigator, Michael Eaton, Principal Investigator, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00000
Record Dates: First submitted 2025-11-24; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Anemia; Iron Deficiency Anemia
Keywords: Anemia; Iron; Transfusion
MeSH Terms: conditions — Anemia; Anemia, Iron-Deficiency | interventions — Therapeutics; sucrosomial iron

STUDY DESIGN:
Intervention Model Description: Randomized 1:1 to IV or oral iron. Hemoglobin and iron study outcomes are planned for the two randomized arms. Participants in the non randomized observational arm will contribute these values only if obtained as part of routine clinical care.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Observer blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- intravenous (IV) iron (Active Comparator): If a participant is to receive IV iron, they will be scheduled to have two infusions, at the URMC Center for Perioperative Medicine (CPM). They will receive the iron through an IV, which is a small plastic tube inserted into a vein in the arm using a needle. This may require that saline water be inserted into the tube to keep the tube from clogging.
  Interventions: Drug: Treatment with intravenous iron
- Sucrosomial Iron (Experimental): If a participant is to receive oral iron capsules, they will be provided with enough capsules to last until the date of surgery and will take 2 capsules every day.
  Interventions: Drug: Treatment with oral sucrosomial iron
- 3rd arm is for data collection only (No Intervention): In addition, 25 patients refusing randomization, but accepting data collection, will be treated as per the standard of care, but will have data collected as for the randomized groups with the exception of no CBC or iron studies will be performed on the day of surgery unless as part of routine care unrelated to study participation.

INTERVENTIONS:
Drug: Treatment with oral sucrosomial iron — blood draw on the day of surgery to check hemoglobin and red blood cell count and iron studies
  Arms: Sucrosomial Iron
Drug: Treatment with intravenous iron — 2 infusions of intravenous iron (ferumoxytol)
  Arms: intravenous (IV) iron

SUMMARY:
50 patients with anemia scheduled for heart surgery or procedures will be randomized to receive either oral sucrosomial iron or standard-of-care intravenous iron before surgery to see if the oral iron is as effective as intravenous iron in increasing the red blood cell count.

DETAILED DESCRIPTION:
Participants will be randomly assigned in a 1 to 1 ratio to one of two treatment groups. One group will receive intravenous (IV) iron, and the other group will receive oral sucrosomial iron.

Participants assigned to the IV iron group will receive two infusions at the University of Rochester Medical Center Center for Perioperative Medicine. Intravenous iron will be administered through a small plastic tube placed into a vein. Saline may be used to maintain the IV line as needed.

Participants assigned to the oral sucrosomial iron group will receive capsules to take at home until the date of surgery, with a dosage of two capsules per day.

All other aspects of perioperative care will follow standard practice. A blood sample for complete blood count and iron studies will be obtained on the day of surgery. This is typically collected when the IV is placed, so an additional needle stick is usually not required.

Randomization applies only to the two treatment arms (intravenous iron and oral sucrosomial iron). The third arm is a non randomized observational cohort for data collection only.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Scheduled for elective cardiac surgical procedures, including:
* Coronary artery bypass graft surgery (CABG)
* Valve procedures
* Aortic root procedures
* Transcatheter aortic valve implantation (TAVI)
* Hemoglobin <12 g/dL and ≥10 g/dL on a complete blood count obtained at the Center for Perioperative Medicine pre operative visit
* Evidence of iron deficiency
* Able to provide informed consent
* Able to understand spoken and written English

Exclusion Criteria:

* Scheduled for cardiac surgery requiring deep hypothermia or circulatory arrest
* Undergoing heart transplantation or ventricular assist device placement
* Lacking capacity to provide informed consent or unable to understand spoken and written English
* Baseline hemoglobin >12 g/dL or <10 g/dL
* Use of anticoagulant medications within 5 days of the Center for Perioperative Medicine visit, or planned initiation of anticoagulant therapy before surgery
* History of hemoglobinopathy
* History of hematologic malignancy
* Bone marrow suppression from non nutritional causes
* Vitamin B12 or folate deficiency
* Known liver disease
* Known kidney disease
* Normal serum iron studies at baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in hemoglobin from baseline to day of surgery or procedure | From the pre operative visit to the day of surgery or procedure, up to approximately eight weeks
  Change in hemoglobin in grams per deciliter from the baseline pre operative complete blood count to the complete blood count obtained on the day of surgery or procedure. Change will be calculated as hemoglobin on the day of surgery minus baseline hemoglobin.

SECONDARY OUTCOMES:
Treatment compliance | From the pre operative visit to the day of surgery or procedure, up to approximately eight weeks
  Proportion of participants who complete the assigned iron treatment. Compliance is defined as receiving both infusions in the intravenous arm and taking the prescribed capsules in the oral arm, based on pill counts and participant reporting.
Proportion of participants receiving any blood transfusion | From the end of surgery or procedure through thirty days post procedure
  Number of participants who receive at least one transfusion of blood products after surgery or procedure
Change in iron study values from baseline to the day of surgery or procedure | From the pre operative visit to the day of surgery or procedure, up to approximately eight weeks
  Change in serum iron, ferritin, and transferrin saturation between baseline and day of surgery
Post operative complications | From the end of surgery or procedure through thirty days
  Number of participants who experience any of the following within thirty days: acute kidney injury, stroke, infection requiring antimicrobial therapy, or death.
Length of intensive care unit stay | 30 days after hospital discharge
  Duration of ICU stay in days, from ICU admission after surgery or procedure until ICU discharge.
Length of hospital stay | 30 days after hospital discharge
  Duration of hospitalization in days, from admission for surgery or procedure until discharge

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Eaton, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Padmanabhan H, Siau K, Curtis J, Ng A, Menon S, Luckraz H, Brookes MJ. Preoperative Anemia and Outcomes in Cardiovascular Surgery: Systematic Review and Meta-Analysis. Ann Thorac Surg. 2019 Dec;108(6):1840-1848. doi: 10.1016/j.athoracsur.2019.04.108. Epub 2019 Jun 21. PMID 31233718
- [Background] Tibi P, McClure RS, Huang J, Baker RA, Fitzgerald D, Mazer CD, Stone M, Chu D, Stammers AH, Dickinson T, Shore-Lesserson L, Ferraris V, Firestone S, Kissoon K, Moffatt-Bruce S. STS/SCA/AmSECT/SABM Update to the Clinical Practice Guidelines on Patient Blood Management. J Extra Corpor Technol. 2021 Jun;53(2):97-124. doi: 10.1182/ject-2100053. No abstract available. PMID 34194077
- [Result] Charytan C, Qunibi W, Bailie GR; Venofer Clinical Studies Group. Comparison of intravenous iron sucrose to oral iron in the treatment of anemic patients with chronic kidney disease not on dialysis. Nephron Clin Pract. 2005;100(3):c55-62. doi: 10.1159/000085049. Epub 2005 Apr 11. PMID 15824508
- [Result] Bertani L, Trico D, Zanzi F, Baiano Svizzero G, Coppini F, de Bortoli N, Bellini M, Antonioli L, Blandizzi C, Marchi S. Oral Sucrosomial Iron Is as Effective as Intravenous Ferric Carboxy-Maltose in Treating Anemia in Patients with Ulcerative Colitis. Nutrients. 2021 Feb 12;13(2):608. doi: 10.3390/nu13020608. PMID 33673371
- [Result] Pierelli L, De Rosa A, Falco M, Papi E, Rondinelli MB, Turani F, Weltert L. Preoperative Sucrosomial Iron Supplementation Increases Haemoglobin and Reduces Transfusion Requirements in Elective Heart Surgery Patients: A Prospective Randomized Study. Surg Technol Int. 2021 Oct 28;39:321-328. doi: 10.52198/21.STI.39.CV1512. PMID 34710946